CLINICAL TRIAL: NCT04489251
Title: Assessment of the TGF-beta Pathway and Micro-RNA in Pediatric Pulmonary Arterial Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Edward Kirkpatrick, Associate Professor, Medical College of Wisconsin
Other Study IDs: 1492809
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; TGF-beta pathway; microRNA
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Exome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum is obtained from the pulmonary artery in patients undergoing a cardiac catheterization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PH subjects: * Pediatric subjects ages 2-17 years
  * Subjects undergoing a clinically indicated cardiac catheterization.
  * Subjects with proven or being evaluated for pulmonary hypertension in WHO classification group 1 or 3†
  * Subjects will be categorized as PAH subjects if they meet the hemodynamic criteria: pulmonary artery pressure >20mmHg, pulmonary vascular resistance index >3 Woods units*m2, and wedge pressures <15mmHg.
  Interventions: Diagnostic Test: Protein Elisa analysis, microRNA analysis, whole exome sequencing
- Control subjects: * Pediatric subjects ages 2-17 years
  * Subjects undergoing a clinically indicated cardiac catheterization.
  * Subjects can be categorized as control subjects if they do not have PH on catheterization and do not meet any exclusion criteria.
  Interventions: Diagnostic Test: Protein Elisa analysis, microRNA analysis, whole exome sequencing

INTERVENTIONS:
Diagnostic Test: Protein Elisa analysis, microRNA analysis, whole exome sequencing — ELISA Testing Procedure: The circulating levels of BMP 2, 4, 6, 7, 9 and 10, together with activin A and TGF-β as well as CHIP will be measured using streptavidin ELISA assays.
  Micro-RNA analysis: From 100µL of plasma, we will prepare small RNA libraries using TruSeq Small RNA Sample Preparation kit (Illumina Inc).
  TGF-B mutation evaluation: Blood from subjects with PH will also be analyzed for known genetic mutations in TGF-B pathway using whole exome sequencing.

SUMMARY:
This is a prospective pilot study to assess the plasma levels of particular proteins involved in the transforming growth factor beta (TGF-β) pathway and its down stream regulators, CHIP, as well as micro RNA molecules in subjects with pulmonary arterial hypertension (PAH) and compare them to control subjects without PAH to see if they can be used as a diagnostic or prognostic marker of PAH and how this compares to other diagnostic biomarkers N-terminal pro-natriuretic peptide (NT Pro-BNP) and C-reactive protein (CRP).

DETAILED DESCRIPTION:
Aim 1: This study will correlate proteins in the TGF- β signaling pathway and micro RNA levels with invasive (catheterization) and non-invasive (echocardiography) measurements of pulmonary artery pressures to assess for the presence and severity of PAH and compare these measurements to the established biomarkers of NT Pro BNP and CRP levels.

Hypothesis 1: Plasma levels of proteins of the TGF-β pathway; bone morphogenic protein (BMP) 2, 4, 6, 7, 9 and 10 along with activin A and TGF-β1 protein as well as CHIP (carboxyl-terminus of Hsp70-intracting protein), an enzyme that regulates the activations and exports of TGF- β to the nucleus will be significantly different in subjects with PH over control subjects.

Hypothesis 2: Plasma levels of proteins in the TGF- β pathway; BMP 2, 4, 6, 7, 9 and 10 along with activin A and TGF-β1 protein as well as CHIP will show better correlation with the presence of PAH and its severity than NT-Pro BNP and CRP levels.

Hypothesis 3: The micro-RNA profiles in plasma will be significantly different in subjects with PAHPH over control subjects.

Aim 2: To correlate protein/micro-RNA levels with clinical status in PAH subjects as assessed by functional status, exercise testing, and PAH drug regimen to determine if they can correlate with disease severity.

Hypothesis 1: Clinical findings in PAH patients will correlate with disease severity and study proteins and micro-RNA levels better than established biomarkers.

Aim 3: To correlate evidence of genetic abnormalities through whole exome sequencing especially in regions known or suspected to cause PAH (e.g. BMPR2, ENG, and ALK1 mutations), within the TGF-β pathway or lung development with the tested protein/micro-RNA levels.

Hypothesis 1: Genetic evaluation of patients with PAH will show abnormalities within the TGF-β pathway or lung development.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects ages 2-17 years
* Subjects undergoing a clinically indicated cardiac catheterization.
* Subjects with proven or being evaluated for pulmonary hypertension in WHO classification group 1 or 3†
* Subjects will be categorized as PAH subjects if they meet the hemodynamic criteria: pulmonary artery pressure >20mmHg, pulmonary vascular resistance index >3 Woods units*m2, and wedge pressures <15mmHg.
* Subjects can be categorized as control subjects if they do not have PH on catheterization and do not meet any exclusion criteria.

Exclusion Criteria:

-

Ages: 2 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Subjects with previously confirmed or suspected to have pulmonary arterial hypertension (PAH) that are undergoing a clinically indicated cardiac catheterization (for diagnostic evaluation) ages 2-17 years are eligible for participation.
  Control subjects undergoing a catheterization as part of an intervention such as atrial septal defect closure or patent ductus arteriosus closure and have a routine right heart catheterization as a part of that procedure and meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of BMP proteins of the TGF-β pathway | One day
  bone morphogenic protein (BMP) 2, 4, 6, 7, 9 and 10 levels will be obtained in PH subjects and will be compared to control subjects in effort to describe how those levels are different in subjects with PH over control subjects. All measured amounts of proteins will be in pg/ml.
Plasma Activin A and TGF-β1 level of the TGF-β pathway | One day
  Activin A and TGF-β1 plasma levels will be obtained in PH subjects and compared to control subjects in effort to describe how those levels are different in subjects with PH over control subjects. All measured amounts will be will be in pg/ml.
Plasma CHIP levels assessment in PH patients and control subjects. | One day
  CHIP (carboxyl-protein terminus of Hsp70-intracting protein) plasma levels will be obtained in PH subjects and compared to control subjects in effort to describe how those levels are different in subjects with PH over control subjects. All measured levels will be in pg/ml

SECONDARY OUTCOMES:
Plasma levels of proteins in the TGF- β pathway and PH disease severity | One day
  BMP 2, 4, 6, 7, 9 and 10 along with activin A and TGF-β1 protein as well as CHIP levels will be correlated with the presence of PAH and its severity and how that compares to the levels of NT-Pro BNP and CRP levels.
MicroRNA levels in PH vs control subjects | One day
  The micro-RNA profiles in plasma will be compared between in subjects with PAH and control subjects.
Clinical findings correlation with study proteins/microRNA | One day
  Clinical findings in PAH patients will be correlated with disease severity and study protein and micro-RNA levels.
Whole exome sequence analysis in PH patients and protein/microRNA levels | One day
  To correlate evidence of genetic abnormalities through whole exome sequencing especially in regions known or suspected to cause PAH (e.g. BMPR2, ENG, and ALK1 mutations), within the TGF-β pathway or lung development with the tested protein/micro-RNA levels.

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Kirkpatrick, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No